CLINICAL TRIAL: NCT05749718
Title: Reliability and Validity of the Turkish Version of the Object Permanence Scale
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Erkan Erol, Assistant Professor, Tokat Gaziosmanpasa University
Other Study IDs: GaziosmanpasaU_Erol_02
Record Dates: First submitted 2023-02-19; First posted 2023-03-01 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Developmental Delay
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is the cultural adaptation of the Object Permanence Scale to Turkish and to examine its validity and reliability. The sample of the study will be 7-16 months old babies with motor developmental delay. Inclusion criteria: 7-16 months of age, sitting for at least 3 seconds but not being able to switch independently between sitting and other positions, and showing at least one developmental delay in the motor development subscale of the Bayley III Developmental Assessment. Evaluations will be done at baseline and after 1 week (retest). Exclusion criteria: Medical complications (eg, severe visual impairment) limiting participation in assessments; autism, down syndrome, or spinal cord injury; diagnosed uncontrolled seizure disorder; or a neurodegenerative disorder.

ELIGIBILITY:
Inclusion Criteria:

* 7-16 months,
* Sitting for at least 3 seconds but unable to independently switch between sitting and other positions
* To show at least one retardation in motor subscale of Bayley III.

Exclusion Criteria:

* Medical complications (eg, severe visual impairment) limiting participation in assessments; autism, down syndrome, or spinal cord injury; diagnosed uncontrolled seizure disorder; or a neurodegenerative disorder

Ages: 7 Months to 16 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants aged 7-16 months with motor developmental delay
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Object Permanence Scale | Baseline
  The minimum score of the Object Permanence Scale is 0, and the maximum score is 10. Higher scores indicate better outcome.
Object Permanence Scale | After 1 week (retest)
  The minimum score of the Object Permanence Scale is 0, and the maximum score is 10. Higher scores indicate better outcome.
The Bayley Scales of Infant and Toddler Development, Third Edition (Bayley-III) motor and cognitive subscales | Baseline
  Cognitive subscale consists of 91 items and Motor subscale consists of 138 items. Items are scored as 1 (done) and 0 (not able to). Higher scores indicate better outcome.
Gross motor function measure sitting subscale | Baseline
  The sitting subscale consists of 20 items. Each item is scored on a 4-point ordinal scale (0-3). Higher scores indicate better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences, Tokat Gaziosmanpaşa University, Tokat Province, Turkey (Türkiye)